CLINICAL TRIAL: NCT03886805
Title: The Effectiveness of Dual-task Training With Variable- and Fixed-priority Instructions on Gait Speed in Community-dwelling Older Adults
Brief Title: The Dual-task Training Under Different Priority Instructions on Gait Speed in Community-dwelling Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pernambuco (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Francis Trombini de Souza, Professor, PhD, University of Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U1111-1229-1346
Record Dates: First submitted 2019-03-12; First posted 2019-03-22 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Gait; Postural Balance

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual task with variable- and fixed-priority instructions (Experimental): Sixty-minute training sessions, 2 times a week for 24 weeks. From the 1st to 12th week the participants were trained under variable-priority instructions (half the session was focused on balance motor task and half the session focused on cognitive task performance). From the 13th to 24th week) the participants performed dual tasks under fixed-priority instructions (simultaneous focus attention on balance and cognitive tasks). The motor tasks were performed in a circuit composed of hula hoops, ropes (in a straight line and zigzag), agility ladder, traffic cones, steps, cardboard box, and other obstacles arranged on the floor (stable surface) or on mattresses (unstable surface), depending on the aiming of each training stage. The cognitive tasks will include activities such as saying fruits, animals, cities, and/or person names started with a specific letter, solving mathematical accounts, singing songs, reciting verses, working memory, among other cognitive tasks.
  Interventions: Other: Dual task with variable- and fixed-priority instructions
- Dual-task with variable-priority instructions (Active Comparator): Sixty-minute training sessions, 2 times a week for 24 weeks (48 sessions). From the 1st to 24th week, the participants were trained under variable-priority instructions, in which they were asked to spend half the session focused on balance (motor task) and half the session focused on cognitive task performance. The motor tasks (gait and postural balance) of this protocol were performed in a circuit composed of hula hoops, ropes (in a straight line and zigzag), agility ladder, traffic cones, steps, cardboard box, and other obstacles arranged on the floor (stable surface) or on mattresses (unstable surface), depending on the aiming of each training stage. The cognitive tasks included activities such as saying fruits, animals, cities, and/or person names started with a specific letter, solving mathematical accounts, singing songs, reciting verses, rescue working memory, among other cognitive tasks.
  Interventions: Other: Dual-task with variable-priority instructions

INTERVENTIONS:
Other: Dual task with variable- and fixed-priority instructions — The participants were asked to perform dual-task activities focused, interchangeable or simultaneously, on balance (motor tasks) and on cognitive tasks performance, according to the instructional priority established by the physical therapist.
  Arms: Dual task with variable- and fixed-priority instructions
Other: Dual-task with variable-priority instructions — The participants were asked to spend half the session focused on balance (motor tasks) and half the session focused on cognitive tasks performance, according to the instructional priority established by the physical therapist.
  Arms: Dual-task with variable-priority instructions

SUMMARY:
This study analyzed the effect of different modalities of dual-task training in the improvement of gait biomechanics, postural balance, falls episodes, executive functioning, and quality of life in community-dwelling older adults. Half of the participants have undertaken a dual-task protocol training with progression from variable-priority to fixed-priority instructions, while the other half have undertaken a dual-task protocol training under variable-priority instructions.

DETAILED DESCRIPTION:
Although dual-task training for improving postural balance is an emerging interest area, the effects of dual tasks and dual-task training on static and dynamic postural stability remain unclear. Even though variable (alternating) instructional priority dual-task training has been shown higher effect than fixed (concurrent) priority dual-task training approach to improving the balance impairments, we must consider in everyday pragmatic situations, motor, and cognitive tasks are often demanded simultaneously and this requires an individual's attention toward an external source of attention while performing a primary task. Then, our rationale for this study is older adults who underwent a training protocol composed of a dual task with variable and fixed instructional priority will achieve better improvements regarding the studied variables in comparison to the group who will be submitted a protocol composed only by dual-task with variable priority training. Therefore, this protocol for a six-month, double-blind, randomized controlled trial with six-month follow-up post-training analyzed whether examine whether a dual-task protocol training with progression from variable priority to fixed priority instructions is effective in improvement of gait biomechanics, postural balance, falls episodes, executive functioning and quality of life in community-dwelling older adults.

ELIGIBILITY:
Inclusion criteria:

* Participants of both sexes
* Age between 60 and 80 years old
* Participants with a score greater or equal to 52 (up to a maximum of 56) in the Berg Balance Scale
* Participants with a score greater or equal to 24 (up to a maximum of 30) in the Mini-mental State Exam
* Participants who are able to walk uninterruptedly for a distance of 10-meter at a self-selected velocity of at least 1.0 m/s without the need from another person, cane or walker

Exclusion criteria:

* Self-report of two or more falls in the last 12 months
* Any contraindication to balance postural training
* Any contraindication to cognitive exercise training
* With self-report of two or more falls in the last 12 months
* Who is participating or have participated, in the last 6 months, in any regular and structured physical exercise program, for 3 or more times per week
* Any chronic health condition, including cardiovascular disease, respiratory disease, stroke, active cancer, neurological or neuromuscular conditions whose exercise is contraindicated
* Any upper or lower limb fracture in the last 6 months
* Evidence of any surgical procedures in the knees, ankles, and hips or muscle damage in the last 6 months
* Uncontrolled diabetes.
* No able to speak and understand the Portuguese language
* Refusal to give informed consent

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
Gait spatiotemporal variables | Post-randomization at week 12
  These variables will be acquired by a couple of inertial sensors attached on participant's feet during walking on a 30-meter flat and level corridor under a single-task (only gait), dual-task under variable- (gait alternating with a cognitive task) and fixed-priority (gait and cognitive task performing simultaneously).
Gait spatiotemporal variables | Post-randomization at week 24
  These variables will be acquired by a couple of inertial sensors attached on participant's feet during walking on a 30-meter flat and level corridor under a single-task (only gait), dual-task under variable- (gait alternating with a cognitive task) and fixed-priority (gait and cognitive task performing simultaneously).
Gait spatiotemporal variables | Post-intervention at week 12
  These variables will be acquired by a couple of inertial sensors attached on participant's feet during walking on a 30-meter flat and level corridor under a single-task (only gait), dual-task under variable- (gait alternating with a cognitive task) and fixed-priority (gait and cognitive task performing simultaneously).
Gait spatiotemporal variables | Post-intervention at week 24
  These variables will be acquired by a couple of inertial sensors attached on participant's feet during walking on a 30-meter flat and level corridor under a single-task (only gait), dual-task under variable- (gait alternating with a cognitive task) and fixed-priority (gait and cognitive task performing simultaneously).

SECONDARY OUTCOMES:
Tri-axial acceleration, angular velocity, and displacement of the body center of mass during gait under single task | Post-randomization at week 12
  These biomechanical variable acquired during gait under single task will be assessed by an inertial sensor fixed on the participant's waist.
Tri-axial acceleration, angular velocity, and displacement of the body center of mass during gait under single task | Post-radomization at week 24
  These biomechanical variable acquired during gait under single task will be assessed by an inertial sensor fixed on the participant's waist.
Tri-axial acceleration, angular velocity, and displacement of the body center of mass during gait under single task | Post-intervention at week 12
  These biomechanical variable acquired during gait under single task will be assessed by an inertial sensor fixed on the participant's waist.
Tri-axial acceleration, angular velocity, and displacement of the body center of mass during gait under single task | Post-intervention at week 24
  These biomechanical variable acquired during gait under single task will be assessed by an inertial sensor fixed on the participant's waist.
Tri-axial acceleration, angular velocity and displacement of the body center of mass during gait under dual-task with variable-priority instruction | Post-randomization at week 12
  These biomechanical variable acquired during gait under dual-task with variable-priority instruction will be assessed by an inertial sensor fixed on the participant's waist.
Tri-axial acceleration, angular velocity and displacement of the body center of mass during gait under dual-task with variable-priority instruction | Post-randomization at week 24
  These biomechanical variable acquired during gait under dual-task with variable-priority instruction will be assessed by an inertial sensor fixed on the participant's waist.
Tri-axial acceleration, angular velocity and displacement of the body center of mass during gait under dual-task with variable-priority instruction | Post-intervention at week 12
  These biomechanical variable acquired during gait under dual-task with variable-priority instruction will be assessed by an inertial sensor fixed on the participant's waist.
Tri-axial acceleration, angular velocity and displacement of the body center of mass during gait under dual-task with variable-priority instruction | Post-intervention at week 24
  These biomechanical variable acquired during gait under dual-task with variable-priority instruction will be assessed by an inertial sensor fixed on the participant's waist.
Tri-axial acceleration, angular velocity and displacement of the body center of mass during gait under dual-task with fixed-priority instruction | Post-randomization at week 12
  These biomechanical variable acquired during gait under dual-task with fixed-priority instruction will be assessed by an inertial sensor fixed on the participant's waist.
Tri-axial acceleration, angular velocity and displacement of the body center of mass during gait under dual-task with fixed-priority instruction | Post-randomization at week 24
  These biomechanical variable acquired during gait under dual-task with fixed-priority instruction will be assessed by an inertial sensor fixed on the participant's waist.
Tri-axial acceleration, angular velocity and displacement of the body center of mass during gait under dual-task with fixed-priority instruction | Post-intervention at week 12
  These biomechanical variable acquired during gait under dual-task with fixed-priority instruction will be assessed by an inertial sensor fixed on the participant's waist.
Tri-axial acceleration, angular velocity and displacement of the body center of mass during gait under dual-task with fixed-priority instruction | Post-intervention at week 24
  These biomechanical variable acquired during gait under dual-task with fixed-priority instruction will be assessed by an inertial sensor fixed on the participant's waist.
Tri-axial acceleration, angular velocity and displacement of the body center of mass during conventional timed up and go test. | Post-randomization at week 12
  These biomechanical variable acquired during conventional timed up and go test will be assessed by an inertial sensor fixed on the participant's waist.
Tri-axial acceleration, angular velocity and displacement of the body center of mass during conventional timed up and go test. | Post-randomization at week 24
  These biomechanical variable acquired during conventional timed up and go test will be assessed by an inertial sensor fixed on the participant's waist.
Tri-axial acceleration, angular velocity and displacement of the body center of mass during conventional timed up and go test. | Post-intervention at week 12
  These biomechanical variable acquired during conventional timed up and go test will be assessed by an inertial sensor fixed on the participant's waist.
Tri-axial acceleration, angular velocity and displacement of the body center of mass during conventional timed up and go test. | Post-intervention at week 24
  These biomechanical variable acquired during conventional timed up and go test will be assessed by an inertial sensor fixed on the participant's waist.
Tri-axial acceleration, angular velocity, and displacement of the body center of mass during manual timed up and go test. | Post-randomization at week 12
  These biomechanical variable acquired during manual timed up and go test will be assessed by an inertial sensor fixed on the participant's waist.
Tri-axial acceleration, angular velocity, and displacement of the body center of mass during manual timed up and go test. | Post-randomization at week 24
  These biomechanical variable acquired during manual timed up and go test will be assessed by an inertial sensor fixed on the participant's waist.
Tri-axial acceleration, angular velocity, and displacement of the body center of mass during manual timed up and go test. | Post-intervention at week 12
  These biomechanical variable acquired during manual timed up and go test will be assessed by an inertial sensor fixed on the participant's waist.
Tri-axial acceleration, angular velocity, and displacement of the body center of mass during manual timed up and go test. | Post-intervention at week 24
  These biomechanical variable acquired during manual timed up and go test will be assessed by an inertial sensor fixed on the participant's waist.
Tri-axial acceleration, angular velocity, and displacement of the body center of mass during cognitive timed up and go test. | Post-randomization at week 12
  These biomechanical variable acquired during cognitive timed up and go test will be assessed by an inertial sensor fixed on the participant's waist.
Tri-axial acceleration, angular velocity, and displacement of the body center of mass during cognitive timed up and go test. | Post-randomization at week 24
  These biomechanical variable acquired during cognitive timed up and go test will be assessed by an inertial sensor fixed on the participant's waist.
Tri-axial acceleration, angular velocity, and displacement of the body center of mass during cognitive timed up and go test. | Post-intervention at week 12
  These biomechanical variable acquired during cognitive timed up and go test will be assessed by an inertial sensor fixed on the participant's waist.
Tri-axial acceleration, angular velocity, and displacement of the body center of mass during cognitive timed up and go test. | Post-intervention at week 24
  These biomechanical variable acquired during cognitive timed up and go test will be assessed by an inertial sensor fixed on the participant's waist.
Tri-axial acceleration, angular velocity, and displacement of the body center of mass during performing the Stroop test in quasi-static standing posture | Post-randomization at week 12
  These biomechanical variable acquired during performing the Stroop test in quasi-static standing posture will be assessed by an inertial sensor fixed on the participant's waist.
Tri-axial acceleration, angular velocity, and displacement of the body center of mass during performing the Stroop test in quasi-static standing posture | Post-randomization at week 24
  These biomechanical variable acquired during performing the Stroop test in quasi-static standing posture will be assessed by an inertial sensor fixed on the participant's waist.
Tri-axial acceleration, angular velocity, and displacement of the body center of mass during performing the Stroop test in quasi-static standing posture | Post-intervention at week 12
  These biomechanical variable acquired during performing the Stroop test in quasi-static standing posture will be assessed by an inertial sensor fixed on the participant's waist.
Tri-axial acceleration, angular velocity, and displacement of the body center of mass during performing the Stroop test in quasi-static standing posture | Post-intervention at week 24
  These biomechanical variable acquired during performing the Stroop test in quasi-static standing posture will be assessed by an inertial sensor fixed on the participant's waist.
Tri-axial acceleration, angular velocity and displacement of the body center of mass during performing the Clinical Test of Sensory Interaction and Balance (CTSIB). | Post-randomization at week 12
  These biomechanical variable acquired during performing the Clinical Test of Sensory Interaction and Balance (CTSIB) will be assessed by an inertial sensor fixed on the participant's waist.
Tri-axial acceleration, angular velocity and displacement of the body center of mass during performing the Clinical Test of Sensory Interaction and Balance (CTSIB). | Post-randomization at week 24
  These biomechanical variable acquired during performing the Clinical Test of Sensory Interaction and Balance (CTSIB) will be assessed by an inertial sensor fixed on the participant's waist.
Tri-axial acceleration, angular velocity and displacement of the body center of mass during performing the Clinical Test of Sensory Interaction and Balance (CTSIB). | Post-intervention at week 12
  These biomechanical variable acquired during performing the Clinical Test of Sensory Interaction and Balance (CTSIB) will be assessed by an inertial sensor fixed on the participant's waist.
Tri-axial acceleration, angular velocity and displacement of the body center of mass during performing the Clinical Test of Sensory Interaction and Balance (CTSIB). | Post-intervention at week 24
  These biomechanical variable acquired during performing the Clinical Test of Sensory Interaction and Balance (CTSIB) will be assessed by an inertial sensor fixed on the participant's waist.
Tri-axial acceleration, angular velocity, and displacement of the body center of mass during performing the Anterior Functional Reach test. | Post-randomization at week 12
  These biomechanical variable acquired during performing the Anterior Functional Reach test will be assessed by an inertial sensor fixed on the participant's waist.
Tri-axial acceleration, angular velocity, and displacement of the body center of mass during performing the Anterior Functional Reach test. | Post-randomization at week 24
  These biomechanical variable acquired during performing the Anterior Functional Reach test will be assessed by an inertial sensor fixed on the participant's waist.
Tri-axial acceleration, angular velocity, and displacement of the body center of mass during performing the Anterior Functional Reach test. | Post-intervention at week 12
  These biomechanical variable acquired during performing the Anterior Functional Reach test will be assessed by an inertial sensor fixed on the participant's waist.
Tri-axial acceleration, angular velocity, and displacement of the body center of mass during performing the Anterior Functional Reach test. | Post-intervention at week 24
  These biomechanical variable acquired during performing the Anterior Functional Reach test will be assessed by an inertial sensor fixed on the participant's waist.
Tri-axial acceleration, angular velocity, and displacement of the body center of mass during performing the Five Times Sit-to-stand test from a chair. | Post-randomization at week 12
  These biomechanical variable acquired during performing the Five Times Sit-to-stand test from a chair will be assessed by an inertial sensor fixed on the participant's waist.
Tri-axial acceleration, angular velocity, and displacement of the body center of mass during performing the Five Times Sit-to-stand test from a chair. | Post-randomization at week 24
  These biomechanical variable acquired during performing the Five Times Sit-to-stand test from a chair will be assessed by an inertial sensor fixed on the participant's waist.
Tri-axial acceleration, angular velocity, and displacement of the body center of mass during performing the Five Times Sit-to-stand test from a chair. | Post-intervention at week 12
  These biomechanical variable acquired during performing the Five Times Sit-to-stand test from a chair will be assessed by an inertial sensor fixed on the participant's waist.
Tri-axial acceleration, angular velocity, and displacement of the body center of mass during performing the Five Times Sit-to-stand test from a chair. | Post-intervention at week 24
  These biomechanical variable acquired during performing the Five Times Sit-to-stand test from a chair will be assessed by an inertial sensor fixed on the participant's waist.
Tri-axial acceleration, angular velocity, and displacement of the body center of mass during performing the Sitting-rising test from the floor. | Post-randomization at week 12
  These biomechanical variable acquired during performing the Sitting-rising test from the floor will be assessed by an inertial sensor fixed on the participant's waist.
Tri-axial acceleration, angular velocity, and displacement of the body center of mass during performing the Sitting-rising test from the floor. | Post-randomization at week 24
  These biomechanical variable acquired during performing the Sitting-rising test from the floor will be assessed by an inertial sensor fixed on the participant's waist.
Tri-axial acceleration, angular velocity, and displacement of the body center of mass during performing the Sitting-rising test from the floor. | Post-intervention at week 12
  These biomechanical variable acquired during performing the Sitting-rising test from the floor will be assessed by an inertial sensor fixed on the participant's waist.
Tri-axial acceleration, angular velocity, and displacement of the body center of mass during performing the Sitting-rising test from the floor. | Post-intervention at week 24
  These biomechanical variable acquired during performing the Sitting-rising test from the floor will be assessed by an inertial sensor fixed on the participant's waist.
Timed Up and Go conventional (TUG conventional) | Post-randomization at week 12
  Test of basic mobility skills analyzed during rising from a chair, walking, turning the obstacle, and sitting again on the chair.
Timed Up and Go conventional (TUG conventional) | Post-randomization at week 24
  Test of basic mobility skills analyzed during rising from a chair, walking, turning the obstacle, and sitting again on the chair.
Timed Up and Go conventional (TUG conventional) | Post-intervention at week 12
  Test of basic mobility skills analyzed during rising from a chair, walking, turning the obstacle, and sitting again on the chair.
Timed Up and Go conventional (TUG conventional) | Post-intervention at week 24
  Test of basic mobility skills analyzed during rising from a chair, walking, turning the obstacle, and sitting again on the chair.
Timed Up and Go manual (TUG manual) | Post-randomization at week 12
  Test of basic mobility skills analyzed during rising from a chair, walking, turning the obstacle, and sitting again on the chair, while the participant carries a dish with a cup on it.
Timed Up and Go manual (TUG manual) | Post-randomization at week 24
  Test of basic mobility skills analyzed during rising from a chair, walking, turning the obstacle, and sitting again on the chair, while the participant carries a dish with a cup on it.
Timed Up and Go manual (TUG manual) | Post-intervention at week 12
  Test of basic mobility skills analyzed during rising from a chair, walking, turning the obstacle, and sitting again on the chair, while the participant carries a dish with a cup on it.
Timed Up and Go manual (TUG manual) | Post-intervention at week 24
  Test of basic mobility skills analyzed during rising from a chair, walking, turning the obstacle, and sitting again on the chair, while the participant carries a dish with a cup on it.
Timed Up and Go cognitive (TUG cognitive) | Post-randomization at week 12
  Test the basic mobility skills analyzed during raising from a chair, walking, bypassing the obstacle, and sitting back in the chair while the participant performs a concurrent cognitive task (solving mathematical subtraction operations).
Timed Up and Go cognitive (TUG cognitive) | Post-randomization at week 24
  Test the basic mobility skills analyzed during raising from a chair, walking, bypassing the obstacle, and sitting back in the chair while the participant performs a concurrent cognitive task (solving mathematical subtraction operations).
Timed Up and Go cognitive (TUG cognitive) | Post-intervention at week 12
  Test the basic mobility skills analyzed during raising from a chair, walking, bypassing the obstacle, and sitting back in the chair while the participant performs a concurrent cognitive task (solving mathematical subtraction operations).
Timed Up and Go cognitive (TUG cognitive) | Post-intervention at week 24
  Test the basic mobility skills analyzed during raising from a chair, walking, bypassing the obstacle, and sitting back in the chair while the participant performs a concurrent cognitive task (solving mathematical subtraction operations).
Postural Balance Test (PBT) | Post-randomization at week 12
  The Postural Balance Test evaluate the static and dynamic balance, in order to verify the typology of motor regulation, i.e. the exteroceptive or visual (six items) and interoceptive or vestibular (eight items), besides the general - proprioceptive information - of the movements.
Postural Balance Test (PBT) | Post-randomization at week 24
  The Postural Balance Test evaluate the static and dynamic balance, in order to verify the typology of motor regulation, i.e. the exteroceptive or visual (six items) and interoceptive or vestibular (eight items), besides the general - proprioceptive information - of the movements.
Postural Balance Test (PBT) | Post-intervention at week 12
  The Postural Balance Test evaluate the static and dynamic balance, in order to verify the typology of motor regulation, i.e. the exteroceptive or visual (six items) and interoceptive or vestibular (eight items), besides the general - proprioceptive information - of the movements.
Postural Balance Test (PBT) | Post-intervention at week 24
  The Postural Balance Test evaluate the static and dynamic balance, in order to verify the typology of motor regulation, i.e. the exteroceptive or visual (six items) and interoceptive or vestibular (eight items), besides the general - proprioceptive information - of the movements.
Clinical Test of Sensory Interaction and Balance (CTSIB) | Post-randomization at week 12
  This test will be used to assess the sensory integration on postural balance during standing on a stable and unstable surface with eyes open and closed.
Clinical Test of Sensory Interaction and Balance (CTSIB) | Post-randomization at week 24
  This test will be used to assess the sensory integration on postural balance during standing on a stable and unstable surface with eyes open and closed.
Clinical Test of Sensory Interaction and Balance (CTSIB) | Post-intervention at week 12
  This test will be used to assess the sensory integration on postural balance during standing on a stable and unstable surface with eyes open and closed.
Clinical Test of Sensory Interaction and Balance (CTSIB) | Post-intervention at week 24
  This test will be used to assess the sensory integration on postural balance during standing on a stable and unstable surface with eyes open and closed.
Stroop test in sit posture | Post-randomization at week 12
  This test will be used to measure a participant's selective attention capacity and skills, as well as his/her processing speed ability in sit posture
Stroop test in sit posture | Post-randomization at week 24
  This test will be used to measure a participant's selective attention capacity and skills, as well as his/her processing speed ability in sit posture
Stroop test in sit posture | Post-intervention at week 12
  This test will be used to measure a participant's selective attention capacity and skills, as well as his/her processing speed ability in sit posture
Stroop test in a quasi-static standing posture | Post-intervention at week 24
  This test will be used to measure a participant's selective attention capacity and skills, as well as his/her processing speed ability in quasi-static standing posture.
Trail making test (TMT) | Post-randomization at week 12
  Trail making test will be used to assess the participants executive abilities, which requires a variety of mental abilities including letter and number recognition mental flexibility, visual scanning, and motor function of upper limbs
Trail making test (TMT) | Post-randomization at week 24
  Trail making test will be used to assess the participants executive abilities, which requires a variety of mental abilities including letter and number recognition mental flexibility, visual scanning, and motor function of upper limbs
Trail making test (TMT) | Post-intervention at week 12
  Trail making test will be used to assess the participants executive abilities, which requires a variety of mental abilities including letter and number recognition mental flexibility, visual scanning, and motor function of upper limbs
Trail making test (TMT) | Post-intervention at week 24
  Trail making test will be used to assess the participants executive abilities, which requires a variety of mental abilities including letter and number recognition mental flexibility, visual scanning, and motor function of upper limbs
Five Times Sit-to-Stand test from a chair | Post-randomization at week 12
  The functional performance of the lower limbs taken to lifting and sitting on a chair for five times. The time will be measured by a stopwatch
Five Times Sit-to-Stand test from a chair | Post-randomization at week 24
  The functional performance of the lower limbs taken to lifting and sitting on a chair for five times. The time will be measured by a stopwatch
Five Times Sit-to-Stand test from a chair | Post-intervention at week 12
  The functional performance of the lower limbs taken to lifting and sitting on a chair for five times. The time will be measured by a stopwatch
Five Times Sit-to-Stand test from a chair | Post-intervention at week 24
  The functional performance of the lower limbs taken to lifting and sitting on a chair for five times. The time will be measured by a stopwatch
Sitting-and-rising test from the floor | Post-randomization at week 12
  Sitting-and-rising test from the floor will be used to quantify how many supports (hands and/or knees or, still, hands on the knees or legs) the individual uses to sit and lift from the floor.
Sitting-and-rising test from the floor | Post-randomization at week 24
  Sitting-and-rising test from the floor will be used to quantify how many supports (hands and/or knees or, still, hands on the knees or legs) the individual uses to sit and lift from the floor.
Sitting-and-rising test from the floor | Post-intervention at week 12
  Sitting-and-rising test from the floor will be used to quantify how many supports (hands and/or knees or, still, hands on the knees or legs) the individual uses to sit and lift from the floor.
Sitting-and-rising test from the floor | Post-intervention at week 24
  Sitting-and-rising test from the floor will be used to quantify how many supports (hands and/or knees or, still, hands on the knees or legs) the individual uses to sit and lift from the floor.
Anterior functional reach test | Post-randomization at week 12
  Anterior functional reach test will be used to determine how far the participants are able to move forward within their stability limit. It is widely used to identify the risk of falling in older adults
Anterior functional reach test | Post-randomization at week 24
  Anterior functional reach test will be used to determine how far the participants are able to move forward within their stability limit. It is widely used to identify the risk of falling in older adults
Anterior functional reach test | Post-intervention at week 12
  Anterior functional reach test will be used to determine how far the participants are able to move forward within their stability limit. It is widely used to identify the risk of falling in older adults
Anterior functional reach test | Post-intervention at week 24
  Anterior functional reach test will be used to determine how far the participants are able to move forward within their stability limit. It is widely used to identify the risk of falling in older adults
Falls Efficacy Scale-International (FES-I) | Post-randomization at week 12
  The 16-item Falls Efficacy Scale-International will be used to measure the participant's fear of falling (the concerns about falling). The sum of all 16 items is considered to compute a total score. The higher the total score achieved by the participant, the higher the concerns about falling.
Falls Efficacy Scale-International (FES-I) | Post-randomization at week 24
  The 16-item Falls Efficacy Scale-International will be used to measure the participant's fear of falling (the concerns about falling). The sum of all 16 items is considered to compute a total score. The higher the total score achieved by the participant, the higher the concerns about falling.
Falls Efficacy Scale-International (FES-I) | Post-intervention at week 12
  The 16-item Falls Efficacy Scale-International will be used to measure the participant's fear of falling (the concerns about falling). The sum of all 16 items is considered to compute a total score. The higher the total score achieved by the participant, the higher the concerns about falling.
Falls Efficacy Scale-International (FES-I) | Post-intervention at week 24
  The 16-item Falls Efficacy Scale-International will be used to measure the participant's fear of falling (the concerns about falling). The sum of all 16 items is considered to compute a total score. The higher the total score achieved by the participant, the higher the concerns about falling.
Activities-specific Balance Confidence (ABC Scale) | Post-randomization at week 12
  The 16-item Activities-specific Balance Confidence Scale will be used to measure the level of balance confidence of the individual during the accomplishment in performing daily activities. The higher the total score achieved by the participant, the higher the level of balance confidence and functioning in daily activities
Activities-specific Balance Confidence (ABC Scale) | Post-randomization at week 24
  The 16-item Activities-specific Balance Confidence Scale will be used to measure the level of balance confidence of the individual during the accomplishment in performing daily activities. The higher the total score achieved by the participant, the higher the level of balance confidence and functioning in daily activities
Activities-specific Balance Confidence (ABC Scale) | Post-intervention at week 12
  The 16-item Activities-specific Balance Confidence Scale will be used to measure the level of balance confidence of the individual during the accomplishment in performing daily activities. The higher the total score achieved by the participant, the higher the level of balance confidence and functioning in daily activities
Activities-specific Balance Confidence (ABC Scale) | Post-intervention at week 24
  The 16-item Activities-specific Balance Confidence Scale will be used to measure the level of balance confidence of the individual during the accomplishment in performing daily activities. The higher the total score achieved by the participant, the higher the level of balance confidence and functioning in daily activities
Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36) | Post-randomization at week 12
  Medical Outcomes Study 36-Item Short-Form Health Survey will be used to evaluate the quality of life of the participants. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability
Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36) | Post-randomization at week 24
  Medical Outcomes Study 36-Item Short-Form Health Survey will be used to evaluate the quality of life of the participants. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability
Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36) | Post-intervention at week 12
  Medical Outcomes Study 36-Item Short-Form Health Survey will be used to evaluate the quality of life of the participants. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability
Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36) | Post-intervention at week 24
  Medical Outcomes Study 36-Item Short-Form Health Survey will be used to evaluate the quality of life of the participants. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability
Short form of the Geriatric Depression Scale (GDS-15) | Post-randomization at week 12
  This 15-item instrument will be used to evaluate the suggestive depression symptoms in the participants. Its items require a yes/no response. Answers indicating depression are in bold and italicized; score one point for each one selected. Each answer "yes" marked with X in questions 3, 4, 6, 8, 9, 10, 12, 14 and 15 or answer "no" noted in questions 1, 5, 7, 11 and 13, computes 1 point. A score of 0 to 5 is normal. A score greater than 5 indicates depression
Short form of the Geriatric Depression Scale (GDS-15) | Post-randomization at week 24
  This 15-item instrument will be used to evaluate the suggestive depression symptoms in the participants. Its items require a yes/no response. Answers indicating depression are in bold and italicized; score one point for each one selected. Each answer "yes" marked with X in questions 3, 4, 6, 8, 9, 10, 12, 14 and 15 or answer "no" noted in questions 1, 5, 7, 11 and 13, computes 1 point. A score of 0 to 5 is normal. A score greater than 5 indicates depression
Short form of the Geriatric Depression Scale (GDS-15) | Post-intervention at week 12
  This 15-item instrument will be used to evaluate the suggestive depression symptoms in the participants. Its items require a yes/no response. Answers indicating depression are in bold and italicized; score one point for each one selected. Each answer "yes" marked with X in questions 3, 4, 6, 8, 9, 10, 12, 14 and 15 or answer "no" noted in questions 1, 5, 7, 11 and 13, computes 1 point. A score of 0 to 5 is normal. A score greater than 5 indicates depression
Short form of the Geriatric Depression Scale (GDS-15) | Post-intervention at week 24
  This 15-item instrument will be used to evaluate the suggestive depression symptoms in the participants. Its items require a yes/no response. Answers indicating depression are in bold and italicized; score one point for each one selected. Each answer "yes" marked with X in questions 3, 4, 6, 8, 9, 10, 12, 14 and 15 or answer "no" noted in questions 1, 5, 7, 11 and 13, computes 1 point. A score of 0 to 5 is normal. A score greater than 5 indicates depression
The falls events | Post-randomization at week 12
  Fall events will be evaluated through a falls diary, delivered monthly by each participant. The participants should note in this diary the day and the fall causes and circumstances.
The falls events | Post-randomization at week 24
  Fall events will be evaluated through a falls diary, delivered monthly by each participant. The participants should note in this diary the day and the fall causes and circumstances.
The falls events | Post-intervention at week 12
  Fall events will be evaluated through a falls diary, delivered monthly by each participant. The participants should note in this diary the day and the fall causes and circumstances.
The falls events | Post-intervention at week 24
  Fall events will be evaluated through a falls diary, delivered monthly by each participant. The participants should note in this diary the day and the fall causes and circumstances.

CONTACTS AND LOCATIONS:
Overall Officials: Francis T de Souza, PhD, Principal Investigator — University of Pernambuco
Locations (1):
- Francis Trombini de Souza, Petrolina, Pernambucano, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Trombini-Souza F, de Maio Nascimento M, da Silva TFA, de Araujo RC, Perracini MR, Sacco ICN. Dual-task training with progression from variable- to fixed-priority instructions versus dual-task training with variable-priority on gait speed in community-dwelling older adults: A protocol for a randomized controlled trial : Variable- and fixed-priority dual-task for older adults. BMC Geriatr. 2020 Feb 22;20(1):76. doi: 10.1186/s12877-020-1479-2. PMID 32087694